CLINICAL TRIAL: NCT06593964
Title: Safety and Efficacy of TACE With Thermosensitive Nanogel Embolic Agent Versus Embosphere for Hepatocellular Carcinoma: A Prospective, Multicenter, Randomized Controlled, Non-inferiority Trial
Brief Title: TACE With Thermosensitive Nanogel Versus Embosphere for HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Dean, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHANCE-2416
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Transarterial Chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE with Thermosensitive Nanogel Embolic Agent (Experimental): Equipment:
  Thermosensitive Nanogel Embolic Agent
  Interventions: Device: Thermosensitive Nanogel Embolic Agent
- TACE with Embosphere Microspheres (Active Comparator): Equipment:
  Embosphere Microspheres
  Interventions: Device: Thermosensitive Nanogel Embolic Agent

INTERVENTIONS:
Device: Thermosensitive Nanogel Embolic Agent — Thermosensitive Nanogel Embolic Agent

SUMMARY:
To verify the safety and efficacy of TACE withThermosensitive Nanogel Embolic Agent for HCC.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled, non-inferiority design trial. Participants who meet the criteria will be randomly assigned into the experimental group or the control group，with a ratio of 1:1. In the experimental group the Thermosensitive Nanogel Embolic Agent will be used in the TACE procedure, while in the control group the Embosphere microspheres will be used. The primary endpoint is disease control rate of the target lesions at 1 month after the last TACE treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese Liver Cancer Staging Scheme, stage IIb-Illa, as well as those with stage Ia-Ila HCC, unsuitable or unwilling to undergo surgical resection, transplantation, or ablation;
2. Liver function status: Child-Pugh A or B
3. Eastern Cooperative Oncology Group score: 0-2 points;
4. With at least one measurable, unembolized liver tumor lesion (1-10 cm) ;
5. Willing to participate in this trial and sign the informed consent.

Exclusion Criteria:

1. The target lesion has been embolized before or require combined with other treatment(s);
2. Diffuse or with extrahepatic metastasis;
3. Coagulation dysfunction (PT prolonged beyond the upper limit of normal for 3 seconds);
4. Severe renal dysfunctions (creatinine clearance rate <30 ml/min);
5. Severe liver dysfunctions (alanine aminotransferase or aspartate aminotransferase exceeding the upper limit of normal by 5 times);
6. Main portal vein was completely occluded and no collateral blood supply was established;
7. With uncorrectable arteriovenous fistula or portal vein fistula;
8. Severe cachexia or hepatic encephalopathy;
9. With active infection;
10. Significant reductions in white blood cells or platelets (white blood cells<3.0x109/L, platelets<50x109/L) that cannot be corrected;
11. Pregnant or lactating women;
12. Difficulty in selective catheterization;
13. With the severe risk of non-target embolization;
14. Severely allergic to contrast agents or the embolic materials;
15. Participating in ongoing trial;
16. Unsuitable judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) | One month after the last TACE
  Probability of target lesion control, evaluated by the investigator and independent image review committee respectively (mRECIST).

SECONDARY OUTCOMES:
Success rate of target lesion embolization | One month after the last TACE
  Success rate of target lesion embolization, evaluated by the investigator and independent image review committee respectively.
Objective response rate (ORR) | One month after the last TACE treatment
  Objective response rate of target lesions, evaluated by the investigator and independent image review committee respectively (mRECIST).
Disease control rate (DCR) | Three and six months after the first TACE
  Probability of target lesion control, evaluated by the investigator and independent image review committee respectively (mRECIST).
Equipment performance evaluation | One month after the first TACE
  (Intraoperative imaging ability, microcatheter delivery capacity) evaluated by the investigator.
Adverse events | Up to 24 months
  Rate of adverse events, evaluated by the investigator (CTACE 5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, M.D., Principal Investigator — Zhongda Hospital
Locations (1):
- Gao-Jun Teng, Nanjing, China

IPD SHARING:
Plan to Share IPD: No